CLINICAL TRIAL: NCT02066610
Title: Effect of Parenteral and Enteral Selenium Supplementation on Trace Mineral Antioxidant Enzyme and Amino Acid Metabolism in Low Birth Weight Infants
Brief Title: Effect of Selenium Supplementation on Trace Mineral Antioxidant Enzyme and Amino Acid Metabolism in Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: AD61
Record Dates: First submitted 2014-02-04; First posted 2014-02-19 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Preterm Infants
MeSH Terms: interventions — Selenium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- PN selenium and formula sodium selenate (Experimental): Parenteral nutrition (PN) with selenium and sodium selenate supplementation of infant formula
  Interventions: Other: selenium and sodium selenate supplementation
- PN selenium and formula sodium selenite (Experimental): Parenteral nutrition (PN) with selenium and sodium selenite supplementation of infant formula
  Interventions: Other: selenium and sodium selenite supplementation
- PN without selenium and formula sodium selenate (Experimental): Parenteral nutrition (PN) without selenium and sodium selenate supplementation of infant formula
  Interventions: Other: Without selenium and sodium selenate supplementation
- PN without selenium and formula sodium selenite (Experimental): Parenteral nutrition (PN) without selenium and sodium selenite supplementation of infant formula
  Interventions: Other: Without selenium and sodium selenite supplementation

INTERVENTIONS:
Other: selenium and sodium selenate supplementation — Parenteral nutrition with selenium and sodium selenate supplementation of infant formula
  Arms: PN selenium and formula sodium selenate
Other: selenium and sodium selenite supplementation — Parenteral nutrition with selenium and sodium selenite supplementation of infant formula
  Arms: PN selenium and formula sodium selenite
Other: Without selenium and sodium selenate supplementation — Parenteral nutrition without selenium and sodium selenate supplementation of infant formula
  Arms: PN without selenium and formula sodium selenate
Other: Without selenium and sodium selenite supplementation — Parenteral nutrition without selenium and sodium selenite supplementation of infant formula
  Arms: PN without selenium and formula sodium selenite

SUMMARY:
The objectives of the study were to assess the serum selenium, zinc, and copper status and plasma and white blood cell antioxidant enzyme activities of low birth weight infants receiving selenium supplemented and non-selenium supplemented parenteral nutrition from initiation of parenteral nutrition until discontinuation of preterm formula or hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* Weight less than 1500 g at birth
* Not capable of receiving enteral feedings prior to 7 days postnatally

Exclusion Criteria:

* Metabolic abnormalities such as inborn errors of metabolism
* Current viral infections
* Enterocolitis confirmed by diagnosis
* Presence of congenital anomalies, severe cardiac disease, liver disease, severe renal and neurological diseases, cholestasis, hemolytic disease and severe gastrointestinal disease
* Evidence of chronic white blood cell disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 1991-03; Primary Completion 1993-06 (Actual); Study Completion 1993-06 (Actual)

PRIMARY OUTCOMES:
Serum Selenium | Change from Baseline to Discharge (~50-60 days)
  4 timepoints include 1) baseline prior to initiation of parenteral nutrition; 2) initiation of enteral nutrition; 3) at discontinuation of parenteral nutrition; 4) at discontinuation of preterm formula/discharge

SECONDARY OUTCOMES:
Weight | Change from study day 1 to study exit (~50-60 days)
  Weight at study day 1, at first enteral feed, at full enteral feeding, and at study exit
Length | Change from study day 1 to study exit (~50-60 days)
  Length at study day 1, at first enteral feed, at full enteral feeding, and at study exit
Head Circumference | Change from study day 1 to study exit (~50-60 days)
  Head circumference at study day 1, at first enteral feed, at full enteral feeding, and at study exit
Intake | Change from study day 1 to study exit (~50-60 days)
  Daily recording of volume and calories from parenteral solutions and study formula consumed
Serum Copper | Change from Baseline to Discharge (~50-60 days)
  4 timepoints include 1) baseline prior to initiation of parenteral nutrition; 2) initiation of enteral nutrition; 3) at discontinuation of parenteral nutrition; 4) at discontinuation of preterm formula/discharge
Serum Zinc | Change from Baseline to Discharge (~50-60 days)
  4 timepoints include 1) baseline prior to initiation of parenteral nutrition; 2) initiation of enteral nutrition; 3) at discontinuation of parenteral nutrition; 4) at discontinuation of preterm formula/discharge
WBC Super oxide dismutase (SOD) activity | Change from Baseline to Discharge (~50-60 days)
  4 timepoints include 1) baseline prior to initiation of parenteral nutrition; 2) initiation of enteral nutrition; 3) at discontinuation of parenteral nutrition; 4) at discontinuation of preterm formula/discharge
Glutathione peroxidase (GSHpx) activity | Change from Baseline to Discharge (~50-60 days)
  4 timepoints include 1) baseline prior to initiation of parenteral nutrition; 2) initiation of enteral nutrition; 3) at discontinuation of parenteral nutrition; 4) at discontinuation of preterm formula/discharge
Plasma GSHpx activity | Change from Baseline to Discharge (~50-60 days)
  4 timepoints include 1) baseline prior to initiation of parenteral nutrition; 2) initiation of enteral nutrition; 3) at discontinuation of parenteral nutrition; 4) at discontinuation of preterm formula/discharge
Plasma Amino Acid Concentrations | Change from Baseline to Discharge (~50-60 days)
  4 timepoints include 1) baseline prior to initiation of parenteral nutrition; 2) initiation of enteral nutrition; 3) at discontinuation of parenteral nutrition; 4) at discontinuation of preterm formula/discharge

CONTACTS AND LOCATIONS:
Overall Officials: Marlene Borschel, Ph.D, Study Chair — Abbott Nutrition
Locations (1):
- Legacy Emanuel Children's Hospital, Portland, Oregon, United States